CLINICAL TRIAL: NCT02480231
Title: Mid-Urethral Sling Tensioning Trial
Acronym: MUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Erin Brennand, Dr., University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB15-0455
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Urinary Stress Incontinence
Keywords: Tension-Free Vaginal Tape; Suburethral Slings; Midurethral Slings; Mid-urethral sling; urinary retention
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Retention | interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Babcock tensioning technique (Active Comparator): Group for whom the retropubic mid-urethral sling was tensioned using a Babcock clamp.
  Interventions: Device: Retropubic Midurethral Sling
- Scissor spacer technique (Active Comparator): Group for whom the retropubic mid-urethral sling was tensioned using a surgical scissor as a spacer.
  Interventions: Device: Retropubic Midurethral Sling

INTERVENTIONS:
Device: Retropubic Midurethral Sling
  Other Names: Tension free Vaginal Tape

SUMMARY:
Prospective randomized clinical trial comparing two methods of intra-operative tensioning of retropubic midurethral slings for stress urinary incontinence. Primary outcome is rate of abnormal bladder function. Secondary outcomes include validated quality of life scores, physical exam findings, and rates of immediate post operative voiding dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Women who have elected for surgical management of symptomatic urinary incontinence
* Ability to read & write in English
* Other prolapse surgery at time of sling placement is allowed
* Must consent to participation in trial

Exclusion Criteria:

* Women with a prior incontinence procedure
* Clinically obvious, but non-symptomatic stress urinary incontinence (latent stress incontinence)
* Declines participation in trial
* Women with existing urinary retention or significant overactive bladder (requiring medication)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2015-09; Primary Completion 2019-04 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Abnormal Bladder Function | 1 year post operative
  Abnormal post-operative bladder function a composite outcome assessed at 12 months after surgery. It is one or more of the following: 1) significantly bothersome stress incontinence or over active bladder symptoms after surgery as measured by questions 1, 2, 3 of the Urogential Distress Inventory (UDI-6) 2) a positive cough stress test in the office, 3) re-treatment for stress urinary incontinence (repeat surgery or pessary use), 4) post-operative urinary retention (presence of self-catheterization at 6 weeks post-operatively or beyond, or therapeutic intervention for retention at any time during the 12 months after, such as pelvic floor physiotherapy, sling lysis, urethrolysis, or sacral nerve stimulation.

SECONDARY OUTCOMES:
Rate of discharge from hospital with on-going need for catheterization | 12 months
Duration of catheterization after surgery | 12 months
Questionnaire scores | 12 months
  standardized questionnaire scores (UDI-6, Incontinence Impact Questionnaire, International Consultation on Incontinence Modular Questionnaire)
Pad test | 12 month
  Standardized 1 hour pad test values
Uroflow parameters | 12 months
  Maximum urine flow rate, post void residual

CONTACTS AND LOCATIONS:
Overall Officials: Erin A Brennand, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Hospital, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brennand EA, Wu G, Houlihan S, Globerman D, Gagnon LH, Birch C, Hyakutake M, Carlson KV, Al-Shankiti H, Robert M, Lazare D, Kim-Fine S; Calgary Women's Pelvic Health Research Group. Two Intraoperative Techniques for Midurethral Sling Tensioning: A Randomized Controlled Trial. Obstet Gynecol. 2020 Sep;136(3):471-481. doi: 10.1097/AOG.0000000000004027. PMID 32769657